CLINICAL TRIAL: NCT02214758
Title: Optimising Nutrition, Oral Health and Medication for Older Home Care Clients
Brief Title: Optimising Nutrition, Oral Health and Medication for Older Home Care Clients (NutOrMed)
Acronym: NutOrMed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Irma Nykänen, PhD, University of Eastern Finland
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RECID84/2012
Record Dates: First submitted 2014-08-04; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Nutrition, Oral Health
Keywords: Home care clients, nutrition, oral health, medication
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dietary counseling (Other)
  Interventions: Other: Nutrition and oral health interventions
- Oral health counseling (Other)
  Interventions: Other: Nutrition and oral health interventions
- nutrition no counseling (No Intervention)
- oral health no counseling (No Intervention)

INTERVENTIONS:
Other: Nutrition and oral health interventions — On the basis of a blood test, Mini Nutritional Assessment, and nutritional anamnesis, the nutritionist developed a plan for individualised nutritional care and discussed with the participant and her/his nurse or family members. If the participants seemed unable to increase the energy and/or protein of their diet, daily complementary dietary drinks were recommended to them. After the dental hygienist interview and oral health examination, the participants in need were targeted for oral health intervention. The intervention included individualised instructions on either dental hygiene, denture hygiene, cleaning of the oral mucosa or for dry mouth. The participants were re-examined six months after the baseline interviews to evaluate the effectiveness of the interventions. Both the intervention and control groups had the same examinations as with the exception of the nutritional and oral health intervention.
  Arms: Dietary counseling; Oral health counseling

SUMMARY:
The aim of the study is to evaluate the impact of six month long nutritional and oral health intervention on nutritional status, oral health, functional performance and hospital admission/costs on older persons using home care services. Additionally, participants are interviewed at home regarding their drugs use and this information will be compared with medication information in electronic patient records.

ELIGIBILITY:
Inclusion Criteria:

* home care clients

Exclusion Criteria:

* under 75 years

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nutritional status on the Mini Nutritional Assessment (MNA) test and s-albumin level at months 6 | Baseline, Month 6
  Using MNA test and s-albumin level test

SECONDARY OUTCOMES:
Change from baseline in oral health status on clinical oral health examination and in-home interview at months 6 | Baseline, Month 6
  Clinical oral health examination included type and location of removable dental prosthesis, examination of the oral mucosa, number and location of teeth, condition of teeth, presence of plaque, gingival bleeding and measurement of periodontal pockets. In-home interview included questions about dental and denture hygiene, a subjective feeling of dry mouth and pain in mouth

OTHER OUTCOMES:
The agreement between medication in-home interview and EMR in baseline | baseline
  A pharmacist recorded each prescription and non-prescription medication and complementary and alternative medicine supplements used regularly, as-needed within a week or in the past on the basis of the interview, medication lists, packages and prescriptions at the baseline. All medications were encoded using the ATC (Anatomic Therapeutic Chemical) classification (WHO). The medication list from the locally used electronic medical record (EMR) was gathered from the same day than in-home interview

CONTACTS AND LOCATIONS:
Overall Officials: Irma Nykänen, PhD, Principal Investigator — University of Eastern Finland

REFERENCES:
- [Derived] Salmi A, Komulainen K, Nihtila A, Tiihonen M, Nykanen I, Hartikainen S, Suominen AL. Eating problems among old home care clients. Clin Exp Dent Res. 2022 Aug;8(4):959-968. doi: 10.1002/cre2.585. Epub 2022 May 8. PMID 35527353
- [Derived] Kaipainen T, Hartikainen S, Tiihonen M, Nykanen I. Effect of individually tailored nutritional counselling on protein and energy intake among older people receiving home care at risk of or having malnutrition: a non-randomised intervention study. BMC Geriatr. 2022 May 4;22(1):391. doi: 10.1186/s12877-022-03088-2. PMID 35505290
- [Derived] Luukkonen A, Tiihonen M, Rissanen T, Hartikainen S, Nykanen I. Orthostatic Hypotension and Associated Factors among Home Care Clients Aged 75 Years or Older - A Population-Based Study. J Nutr Health Aging. 2018;22(1):154-158. doi: 10.1007/s12603-017-0953-9. PMID 29300435
- [Derived] Miettinen M, Tiihonen M, Hartikainen S, Nykanen I. Prevalence and risk factors of frailty among home care clients. BMC Geriatr. 2017 Nov 17;17(1):266. doi: 10.1186/s12877-017-0660-8. PMID 29149866
- [Derived] Tiihonen M, Hartikainen S, Nykanen I. Chair rise capacity and associated factors in older home-care clients. Scand J Public Health. 2018 Nov;46(7):699-703. doi: 10.1177/1403494817718072. Epub 2017 Jul 12. PMID 28699419
- [Derived] Polonen S, Tiihonen M, Hartikainen S, Nykanen I. Individually Tailored Dietary Counseling among Old Home Care Clients - Effects on Nutritional Status. J Nutr Health Aging. 2017;21(5):567-572. doi: 10.1007/s12603-016-0815-x. PMID 28448088